CLINICAL TRIAL: NCT01797705
Title: Revised Algorithm for Next Generation DeVilbiss AutoAdjust CPAP
Brief Title: Revised Algorithm for Next Generation DeVilbiss Healthcare AutoAdjust Continuous Positive Airway Pressure (CPAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DeVilbiss Healthcare LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DHC-002
Record Dates: First submitted 2013-01-08; First posted 2013-02-22 (Estimated); Results first posted 2015-04-28 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Experimental): All subjects underwent a sleep study with DeVilbiss AutoAdjust CPAP with revised algorithm simultaneously with hand-scored PSG.
  Interventions: Device: DeVilbiss AutoAdjust CPAP with revised algorithm

INTERVENTIONS:
Device: DeVilbiss AutoAdjust CPAP with revised algorithm — Subjects attended a one-night polysomnogram (PSG) titration study. DeVilbiss AutoAdjust CPAP with a revised algorithm was compared to hand-scored PSG to determine whether the machine results were equivalent to hand scores. Each subject acted as their own control for assessing accuracy of sleep event analysis and prescribed CPAP pressure.

SUMMARY:
The purpose of this protocol is to improve the current FDA-approved continuous positive pressure auto-titration algorithm, including treatment precision, residual disease detection characteristics and phenotyping with the DeVilbiss brand AutoAdjust CPAP device.

ELIGIBILITY:
Inclusion Criteria:

* Apnea hypopnea index ≥ 15 / hour of sleep on the diagnostic polysomnogram, or diagnostic component of a split night polysomnogram
* Sleep efficiency reported on CPAP titration night PSG should be > 78%
* Diagnosis of moderate to severe obstructive sleep apnea (AHI ≥15) or central/complex sleep apnea
* On stable CPAP or APAP [Automatic Positive Airway Pressure] therapy, with compliant use averaging 4 or more hours nightly
* Age 21-75 years
* Predominately central sleep apnea for up to 10 subjects only
* Willingness to give written informed consent and ability to adhere to visit schedule

Exclusion Criteria:

Diagnosis of mild sleep apnea

* CPAP naïve patients
* Co-morbid conditions which render participation to be at risk. These may include patients with congestive heart failure, COPD [Chronic Obstructive Pulmonary Disease] or psychiatric illness
* Allergies to mask materials
* Evidence of another primary sleep disorder
* Evidence of arousing periodic limb movements during titration
* Contraindications as listed on product labeling
* Pregnant
* Currently diagnosed with depression if symptomatic
* Deemed medically unsuitable by investigator
* Evidence of any type of infection or treatment of an infectious condition during the period of research participation
* Have a bi-level requirement, or prescribed a bi-level therapy device
* CPAP pressure >15cmH2O
* Subjects with tracheotomy
* Uncontrolled hypertension
* Require supplemental oxygen
* Stimulants, major tranquillizers or antipsychotics
* Restless Leg Syndrome or Periodic Leg Movement Index of > 5 per hour

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- NeuroCare, Inc., Newton, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: All enrolled subjects
Period: Overall Study
Arm/Group | All Subjects
Started | 33
Completed | 28
Not Completed | 5
Not completed — Equipment anomalies during sleep studies | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Subjects completing the study with evaluable results
Groups:
- All Evaluable Subjects: All subjects completing the one-night sleep study with evaluable results.
Arm/Group | All Evaluable Subjects
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 16
Apnea Type at Enrollment [Number; unit: participants] — Number of participants with obstructive vs central apnea at enrollment
  participants
    Obstructive Sleep Apnea | 26
    Central Sleep Apnea | 2

OUTCOME MEASURES:

1. Primary Outcome: % Agreement Between Reviewer and Machine Pressure Settings During Sleep Study
Description: The primary objective for the study was demonstrating effectiveness of therapy provided by the DeVilbiss AutoAdjust device as reported by the expert human reviewer. The primary endpoint was that expert human reviewer should agree with pressure changes made by the machine during each 20-minute epoch at least 80% of the time. Expert human reviewer reviewed each study and made a determination at 20-minute time points, in context of REM/NON-REM sleep and supine/non-supine positions, marking the machine pressure response with an "agree" or "disagree." Pressure changes might show no change, increase or decrease during the 20-minute epoch.
Time Frame: 1 night
Population: Subjects completing the study with evaluable results
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Arm/Group | All Evaluable Subjects
Number analyzed (Participants) | 28
percentage of agreement | 92.2 [89.9 to 94.2]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for the period from patient's enrollment in the study up to termination (the morning following the one-night sleep study).
Description: Adverse events were assessed per a list of probable events associated with use of CPAP equipment. There were no adverse events for the analysis population.
Groups:
- Evaluable Subjects: All subjects completing the one-night sleep study with evaluable results.
Arm/Group | Evaluable Subjects
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No